CLINICAL TRIAL: NCT00721513
Title: Phase II Study to Evaluate the Efficacy and Toxicity of Multimodality Treatment With Induction Taxotere/Cisplatin?5-FU (TPF) Chemotherapy Followed by Concomitant Cetuximab and Radiation Therapy in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Docetaxel, Cisplatin, and Fluorouracil Followed By Cetuximab and Radiation Therapy in Treating Patients With Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005784; P30CA012197 (NIH); CCCWFU-60108; CCCWFU-IRB- IRB00005784; SANOFI-AVENTIS-CCCWFU-60108
Record Dates: First submitted 2008-07-23; First posted 2008-07-24 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Docetaxel; Fluorouracil; Magnetic Resonance Spectroscopy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TPFChemotherapy + Concomitant Cetuximab & RT (Experimental): Taxotere/Cisplatinum/5-Fluorouracil (TPF) Chemotherapy Followed by Concomitant Cetuximab & Radiation Therapy
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: docetaxel; Drug: fluorouracil; Procedure: computed tomography; Procedure: positron emission tomography; Procedure: quality-of-life assessment; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin
Drug: docetaxel
Drug: fluorouracil
Procedure: computed tomography
Procedure: positron emission tomography
Procedure: quality-of-life assessment
Radiation: 3-dimensional conformal radiation therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, cisplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with cetuximab and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel, cisplatin, and fluorouracil together with cetuximab and radiation therapy works in treating patients with locally advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the progression-free survival of patients with locally advanced squamous cell carcinoma of the head and neck treated with induction chemotherapy comprising docetaxel, cisplatin, and fluorouracil followed by concurrent cetuximab and radiotherapy.

Secondary

* Assess the objective response rate in patients treated with this regimen.
* Assess the best overall response rate, overall survival, local-regional control, and distant failure in patients treated with this regimen.
* Assess the acute and long-term toxicity associated with this regimen in these patients.
* Assess quality of life and swallowing in patients treated with this regimen.
* Determine the accuracy of PET/CT scan in evaluating objective response; in detecting residual disease at primary sites and nodes; in guiding the recommendation for salvage surgery or for neck dissection; and in early detection of recurrent or metastatic disease.

OUTLINE: Patients are stratified according to nodal status (N2b-c or N3 vs N0-2a), tumor characteristics of invasiveness (present vs absent), human papilloma virus (HPV) status (positive vs negative), and primary tumor site (hypopharynx vs larynx vs oropharynx).

Patients receive induction chemotherapy comprising docetaxel IV over 1 hour and cisplatin IV over 1 hour on day 1 and fluorouracil IV continuously on days 1-4. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-4 weeks after completion of induction chemotherapy, patients receive cetuximab IV once weekly for 7 weeks. Beginning 1 week after the first dose of cetuximab, patients undergo concurrent intensity-modulated radiotherapy or conventional 3-dimensional radiotherapy once or twice daily 5-6 days a week for up to 6 weeks. Patients with persistent disease undergo salvage resection of the primary tumor and/or neck dissection approximately 3 months after the completion of radiotherapy.

Patients undergo quality of life and swallowing evaluations periodically.

Patients undergo PET/CT scan at baseline, before beginning radiotherapy, at 6-8 weeks after completion of study treatment, every 6 months for 5 years, and then annually thereafter.

After completion of study treatment, patients are followed at 4 and 8 weeks, every 2 months for 2 years, every 3 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion:

* Histologically confirmed (from primary lesion and/or lymph nodes) squamous cell carcinoma (SCC) of the head and neck, including the following subtypes:

  * Oropharynx
  * Hypopharynx
  * Larynx
* Primary site of tumor must not include any of the following:

  * Nasopharynx
  * Sinuses
  * Salivary glands
* Stage III or IV disease that is unresectable (oropharynx, larynx, or hypopharynx) OR that is resectable with organ-sparing goal (oropharynx or hypopharynx)
* Measurable disease by CT scan or MRI
* No definitive evidence of distant metastasis
* ECOG performance status 0-1
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 8 g/dL
* Total bilirubin ≤ normal

  * Except in the case where the elevated total bilirubin is not a sign of liver disease (i.e., Gilbert syndrome), in which case a total bilirubin ≤ 2 times upper limit of normal (ULN) is allowed provided direct bilirubin is ≤ ULN
* AST, ALT, and alkaline phosphate (AP) meeting the following criteria:

  * AP normal AND AST or ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal
* Creatinine ≤ 1.5 mg/dL
* Negative pregnancy test (for women of childbearing potential)
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* Willing to undergo laryngoscopy with biopsy of residual tumor at primary site (as part of a comprehensive evaluation of tumor response after completion of the induction chemotherapy portion of study treatment)

Exclusion:

* History of severe hypersensitivity reaction to docetaxel or to other drugs formulated with polysorbate 80
* Other invasive malignancy within the past 3 years, except nonmelanoma skin cancer
* Prior allergic reaction to the study drug(s)
* Concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Psychiatric illness/social situation that would limit compliance with study requirements
  * Significant history of uncontrolled cardiac disease, including any of the following:

    * Uncontrolled hypertension
    * Unstable angina
    * Myocardial infarction within the past 6 months
    * Uncontrolled congestive heart failure
    * Cardiomyopathy with decreased left ventricular ejection fraction (i.e., LVEF < 45%)
* Uncontrolled condition that, in the opinion of the investigator, would interfere in the safe and timely completion of study procedures
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on screening chest CT scan
* HIV positivity
* Pregnant or nursing
* Prior chemotherapy for the study cancer
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiotherapy fields
* Prior chemotherapy, biological therapy, or hormone therapy within the last one year
* Prior initial surgical treatment, except diagnostic biopsy of the primary site or nodal sampling of neck disease
* Prior radical or modified neck dissection
* Prior therapy that specifically and directly targets the EGFR pathway
* Concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Porosnicu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TPFChemotherapy + Concomitant Cetuximab & RT: Taxotere/Cisplatinum/5-Fluorouracil (TPF) Chemotherapy Followed by Concomitant Cetuximab & Radiation Therapy
  cetuximab
  cisplatin
  docetaxel
  fluorouracil
  computed tomography
  positron emission tomography
  quality-of-life assessment
  3-dimensional conformal radiation therapy
  intensity-modulated radiation therapy
Period: Overall Study
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (6.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Time Frame: up to 2 years
Measure: Median (Standard Error); unit: months
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 20
months | 54.2 (0.5)

2. Secondary Outcome: Objective Response Rate
Description: Will be measured by CT scan /MRI of the head and neck with corroborative results of direct biopsy of any residual tumor at primary site.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 20
Participants
  Complete response | 5
  Partial response | 10
  Stable disease | 1
  Progression of disease | 4

3. Secondary Outcome: Best Overall Response Rate
Description: Defined as rate of complete and partial responses (at least 30% decrease in the sum of the longest diameter of target lesions), measured by CT scan or MRI of the head and neck after completion of multimodality treatment with induction TPF (Docetaxel, cisplatin and fluorouracil) chemotherapy followed by combined ERT. We will use RECIST (Response Evaluation Criteria In Solid Tumors) (Therasse et al, 2000) for evaluation of response.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 20
Participants
  Complete response | 5
  Partial response | 10
  Progression of disease | 4
  Stable disease | 1

4. Secondary Outcome: Overall Survival
Time Frame: up to 2 years
Measure: Median (Standard Error); unit: months
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 20
months | 53.6 (0.5)

5. Secondary Outcome: Number of Participants With Distant Metastasis
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 20
Participants | 3

6. Secondary Outcome: Quality of Life - Functional Assessment of Cancer Therapy - General (FACT-G)
Description: Four subscales: physical well-being (PWB; 7-items, score range 0-28), social/family well-being (SWB; 7-items, score range 0-28), emotional well-being (EWB; 6-items, score range 0-24), and functional well-being (FWB; 7-items, score range 0-28). Items are rated on a five-point scale: 0-"not at all", 1- "a little bit", 2-"somewhat", 3- "quite a bit" and 4-"very much". Overall quality of life is the sum of the core items of the FACT-G possible range of 0-108 points. The higher the score the better the quality life. This interval includes 0, we will conclude that there is not conclusive statistical evidence that there is an improvement or worsening. If the interval does not include 0 we can determine whether there was a significant improvement (or worsening) depending on which side of the 0 the interval is on. The total outcome index score (possible range 0-108 points) is the sum of the physical and functional well being and additional concerns categories from the FACT-G.
Time Frame: Baseline, pre-radiation therapy and post-radiation therapy, up to 2 years
Population: This data was not collected on all participants.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 16
Score on a scale
  Baseline - Physical Well-Being | 17.21 [13.14 to 21.25]
  Baseline - Social/Family Well-Being | 23.66 [21.40 to 25.92]
  Baseline - Emotional Well-Being | 17.00 [14.30 to 19.70]
  Baseline Functional Well-Being | 17.48 [14.00 to 20.95]
  Baseline Total Fact-G Score | 75.35 [65.84 to 84.86]
  Baseline Additional Concerns | 23.25 [18.67 to 27.83]
  Total Outcome Index Score - Baseline | 57.94 [48.05 to 67.82]
  Pre-RT Physical Well-Being: number analyzed (Participants) | 9
  Pre-RT Physical Well-Being | 15.56 [10.59 to 20.52]
  Pre-RT Social/Family Well-Being: number analyzed (Participants) | 10
  Pre-RT Social/Family Well-Being | 23.90 [21.24 to 26.56]
  Pre-RT Emotional Well-Being: number analyzed (Participants) | 10
  Pre-RT Emotional Well-Being | 18.80 [15.55 to 22.05]
  Pre-RT Functional Well-Being: number analyzed (Participants) | 10
  Pre-RT Functional Well-Being | 15.63 [11.55 to 19.72]
  Pre-RT Total Fact-G Score: number analyzed (Participants) | 9
  Pre-RT Total Fact-G Score | 72.00 [59.13 to 84.87]
  Pre-RT Additional Concerns: number analyzed (Participants) | 9
  Pre-RT Additional Concerns | 25.44 [20.43 to 30.46]
  Total Outcome Index Score - Pre-RT: number analyzed (Participants) | 9
  Total Outcome Index Score - Pre-RT | 55.78 [44.79 to 66.76]
  Post-RT Social/Family Well-Being: number analyzed (Participants) | 12
  Post-RT Social/Family Well-Being | 23.80 [20.74 to 26.86]
  Post-RT Physical Well-Being: number analyzed (Participants) | 12
  Post-RT Physical Well-Being | 16.42 [11.08 to 21.75]
  Post-RT Emotional Well-Bein: number analyzed (Participants) | 12
  Post-RT Emotional Well-Bein | 18.93 [16.10 to 21.77]
  Post-RT Functional Well-Being: number analyzed (Participants) | 12
  Post-RT Functional Well-Being | 15.92 [10.72 to 21.11]
  Post-RT FACT-G Total Score: number analyzed (Participants) | 12
  Post-RT FACT-G Total Score | 75.07 [60.17 to 89.97]
  Post-RT Additional Concerns: number analyzed (Participants) | 12
  Post-RT Additional Concerns | 21.28 [15.40 to 27.16]
  Total Outcome Index Score - Post- RT: number analyzed (Participants) | 12
  Total Outcome Index Score - Post- RT | 50.00 [-22.63 to 122.63]

7. Secondary Outcome: Number of Participants With Local-Regional Control
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 20
Participants | 20

8. Secondary Outcome: Performance Status Scale for Head and Neck Cancer
Description: Consists of assessment of three functions (subscales): Normalcy of diet, eating in public, and understandability of speech. The interviewer rates the patient on each scale based on the patient's responses to targeted questions. Scores range from 0-100 (Full performance (100 score), moderate or severe impairment (≤ 50 score)). The higher the score, the better the ability of the patient to function.
Time Frame: Baseline, pre-radiation therapy and post-radiation therapy, up to 2 years
Population: Data was not collected for all participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 16
Score on a scale
  Baseline Performance Status for Eating: number analyzed (Participants) | 10
  Baseline Performance Status for Eating | 82.50 (26.48)
  Baseline Performance Status for Speech: number analyzed (Participants) | 10
  Baseline Performance Status for Speech | 95.00 (10.54)
  Baseline Performance Status for Diet: number analyzed (Participants) | 9
  Baseline Performance Status for Diet | 84.44 (20.07)
  Pre-RT Performance Status for Eating: number analyzed (Participants) | 6
  Pre-RT Performance Status for Eating | 45.83 (51.03)
  Pre-RT Performance Status for Speech: number analyzed (Participants) | 6
  Pre-RT Performance Status for Speech | 100.00 (0.00)
  Pre-RT Performance Status for Diet: number analyzed (Participants) | 6
  Pre-RT Performance Status for Diet | 41.67 (49.16)
  Post-RT Performance Status for Eating: number analyzed (Participants) | 4
  Post-RT Performance Status for Eating | 50.00 (45.64)
  Post-RT Performance Status for Speech: number analyzed (Participants) | 4
  Post-RT Performance Status for Speech | 93.75 (12.50)
  Post-RT Performance Status for Diet: number analyzed (Participants) | 4
  Post-RT Performance Status for Diet | 40.00 (45.46)

9. Secondary Outcome: MD Anderson Dysphagia Inventory
Description: The MD Anderson Dysphasia Inventory (MDADI) is a survey specifically designed to assess dysphasia. It contains 20 questions directly addressing the swallowing function and several other general questions. The questionnaire asks for participants views about their swallowing ability at baseline, pre-radiation therapy and post-radiation therapy. All questions except for E7 and F2: Strongly Agree = 1 point, Agree = 2 points, No Opinion = 3 points, Disagree = 4 points, Strongly Disagree. E7 and F2: Strongly agree = 5 points, Agree = 4 points, no opinion = 3 points, disagree = 2 points, strongly disagree = 1 point. Scores range from 20 (extremely low-functioning) to 100 (high-functioning).
Time Frame: Baseline, pre-radiation therapy and post-radiation therapy, up to 2 years
Population: Data was not collected on all participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
Number analyzed (Participants) | 10
Score on a scale
  Baseline Global Score | 56.00 (32.39)
  Baseline Emotion Score: number analyzed (Participants) | 9
  Baseline Emotion Score | 71.48 (16.68)
  Baseline Function Score: number analyzed (Participants) | 9
  Baseline Function Score | 75.56 (20.34)
  Baseline Physical Score | 68.00 (22.94)
  Pre-RT Global Score: number analyzed (Participants) | 5
  Pre-RT Global Score | 88.00 (26.83)
  Pre-RT Emotion Score: number analyzed (Participants) | 5
  Pre-RT Emotion Score | 83.07 (6.35)
  Pre-RT Function Score: number analyzed (Participants) | 5
  Pre-RT Function Score | 76.80 (9.96)
  Pre-RT Physical Score: number analyzed (Participants) | 5
  Pre-RT Physical Score | 86.00 (19.89)
  Post-RT Global Score: number analyzed (Participants) | 8
  Post-RT Global Score | 62.50 (36.15)
  Post-RT Emotion Score: number analyzed (Participants) | 8
  Post-RT Emotion Score | 67.08 (17.59)
  Post-RT Function Score: number analyzed (Participants) | 7
  Post-RT Function Score | 58.29 (26.62)
  Post-RT Physical Score: number analyzed (Participants) | 8
  Post-RT Physical Score | 67.81 (26.47)

ADVERSE EVENTS:
Time Frame: Up to 2 years after completion of treatment
Arm/Group | TPFChemotherapy + Concomitant Cetuximab & RT
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 20/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPFChemotherapy + Concomitant Cetuximab & RT (N=20)
Low WBC (Investigations) | 7 (7)
low Platelets (Investigations) | 1 (1)
Low Hemoglobin (Investigations) | 10 (10)
Vomiting (Gastrointestinal disorders) | 1 (1)
Anorexia (General disorders) | 4 (4)
Low ANC (Investigations) | 9 (9)
Fatigue (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
hyperglycemia (Investigations) | 3 (3)
hypocalcemia (Investigations) | 2 (2)
hypomagnesemia (Investigations) | 1 (1)
hyponatremia (Investigations) | 13 (13)
hypokalemia (Investigations) | 9 (9)
Bicarbonate serum-low (Investigations) | 1 (1)
hyperbilirubinemia (Investigations) | 1 (1)
hypophosphatemia (Investigations) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
hypermagnesemia (Investigations) | 1 (1)
hyperkalemia (Investigations) | 2 (2)
Dysphagia (General disorders) | 4 (4)
Fever without neutropenia (General disorders) | 1 (1)
Febrile neutropenia (Investigations) | 1 (1)
Dry mouth (General disorders) | 1 (1)
Hypoxia (Investigations) | 1 (1)
Dehydration (General disorders) | 3 (3)
Pain: Abdomen (General disorders) | 1 (1)
Acidosis (Investigations) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain: Back (General disorders) | 1 (1)
Colitis (Infections and infestations) | 1 (1)
Death not associated with any term (General disorders) | 1 (1)
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphopenia (Investigations) | 17 (17)
Pain Oral cavity (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Rash: dermatitis associated with radiation: Chemoradiation (Skin and subcutaneous tissue disorders) | 1 (1)
Dental problems (General disorders) | 5 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils: Pleura (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: Abdomen (Infections and infestations) | 1 (1)
Pain: Tumor pain (General disorders) | 1 (1)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 6 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPFChemotherapy + Concomitant Cetuximab & RT (N=20)
Low WBC (Investigations) | 10 (10)
low Platelets (Investigations) | 14 (14)
Low Hemoglobin (Investigations) | 10 (10)
Nausea (Gastrointestinal disorders) | 18 (18)
Vomiting (Gastrointestinal disorders) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Anorexia (General disorders) | 7 (7)
Gastrointestinal - Other (General disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 9 (9)
Creatinine (Investigations) | 6 (6)
Proteinuria (Investigations) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypertension (General disorders) | 5 (5)
Hypotension (Cardiac disorders) | 8 (8)
Neuropathy: sensory (Cardiac disorders) | 5 (5)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Low ANC (Investigations) | 2 (2)
Pain (General disorders) | 1 (1)
Dizziness (General disorders) | 6 (6)
Taste alteration (General disorders) | 6 (6)
Insomnia (General disorders) | 3 (3)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Rigors/chills (General disorders) | 6 (6)
Sweating (General disorders) | 2 (2)
Fatigue (General disorders) | 16 (16)
Weight loss (General disorders) | 8 (8)
hyperglycemia (Investigations) | 17 (17)
hypoglycemia (Investigations) | 1 (1)
hypercalcemia (Investigations) | 1 (1)
hypocalcemia (Investigations) | 18 (18)
hypomagnesemia (Investigations) | 16 (16)
hyponatremia (Investigations) | 7 (7)
hypokalemia (Investigations) | 5 (5)
Bicarbonate serum-low (Investigations) | 5 (5)
hypoalbuminemia (Investigations) | 18 (18)
hyperbilirubinemia (Investigations) | 5 (5)
serum glutamic pyruvic transaminase (Investigations) | 6 (6)
hypophosphatemia (Investigations) | 9 (10)
Constipation (Gastrointestinal disorders) | 15 (15)
Pain: Head/headache (General disorders) | 9 (9)
serum glutamic oxaloacetic transaminase (Investigations) | 6 (6)
hypermagnesemia (Investigations) | 3 (3)
hyperkalemia (Investigations) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1)
Ocular/Visual - Other (Eye disorders) | 1 (1)
Dysphagia (General disorders) | 13 (13)
Fever without neutropenia (General disorders) | 5 (5)
Urinary frequency/urgency (General disorders) | 2 (2)
Infection - Other (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Edema: head and neck (Vascular disorders) | 3 (3)
Edema: limb (Vascular disorders) | 6 (6)
Edema: viscera (Vascular disorders) | 1 (1)
Heartburn/dyspepsia (General disorders) | 4 (4)
Dry mouth (General disorders) | 7 (7)
Dehydration (General disorders) | 5 (5)
Confusion (General disorders) | 1 (1)
Pruritus/itching (General disorders) | 3 (3)
Anxiety (General disorders) | 4 (4)
Depression (General disorders) | 5 (5)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10 (10)
Distension bloating, abdominal (General disorders) | 1 (1)
Pain: Abdomen (General disorders) | 8 (9)
Acidosis (Investigations) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Partial Thromboplastin Time (Investigations) | 5 (5)
Pain: Joint (General disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pain: Back (General disorders) | 3 (3)
Pain: Bone (General disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: Bronchus (Infections and infestations) | 1 (1)
Bronchospasm wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain: Chest/thorax (General disorders) | 1 (1)
Pain: Chest wall (General disorders) | 2 (2)
Colitis infectious (Infections and infestations) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Wound complication, non-infectious (General disorders) | 2 (2)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 (5)
Rash: dermatitis associated with radiation (Skin and subcutaneous tissue disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Hemorrhage respiratory (Vascular disorders) | 1 (1)
Extrapyramidal/involuntary movement/restlessness (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (4)
Flushing (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
gamma-Glutamyl transpeptidase (Investigations) | 2 (2)
Pain: Oral-gums (General disorders) | 1 (1)
Glomerular filtration rate (Investigations) | 5 (5)
Cholesterol, serum-high (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (2)
hypertriglyceridemia (Investigations) | 1 (1)
functional obstruction of bowel (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: Kidney (Infections and infestations) | 1 (1)
Voice changes (General disorders) | 2 (2)
Lymphopenia (Investigations) | 3 (3)
Memory impairment (General disorders) | 1 (1)
Muscle weakness (General disorders) | 7 (7)
Pain: Muscle (General disorders) | 1 (1)
Nail changes (General disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils: Mucosa (Infections and infestations) | 1 (1)
Pain: Neck (General disorders) | 7 (8)
infection associated with Lymphopenia (Infections and infestations) | 1 (1)
Pain Oral cavity (General disorders) | 5 (6)
Pain: Extremity-limb (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Pain: Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pain: Throat/pharynx/larynx (General disorders) | 10 (10)
Pain: Pleura (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Rash: dermatitis associated with radiation: Chemoradiation (Skin and subcutaneous tissue disorders) | 6 (6)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 3 (3)
Salivary gland changes/saliva (General disorders) | 6 (6)
Supraventricular and nodal arrhythmia: Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Pain: Dental/teeth/peridontal (General disorders) | 1 (1)
Neuropathy: cranial: CN V Motor-jaw muscles; Sensory-facial (General disorders) | 2 (2)
Trismus (difficulty, restriction or pain when opening mouth) (General disorders) | 4 (4)
Pain: Urethra (General disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (1)
Hemorrhage GU: Urinary (Vascular disorders) | 2 (2)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 1 (1)
Cytokine release syndrome/acute infusion reaction (General disorders) | 1 (1)
Pain: Anus (General disorders) | 1 (1)
Pain: Tumor pain (General disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils: Foreign body (Infections and infestations) | 1 (1)
Mucositis/stomatitis Oral cavity (Infections and infestations) | 11 (11)
Hemorrhage pulmonary/upper respiratory (Vascular disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils: Wound (Infections and infestations) | 1 (1)
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower (Musculoskeletal and connective tissue disorders) | 2 (2)
Neuropathy: cranial: CN VIII Hearing and balance (Ear and labyrinth disorders) | 2 (2)
Pain: External ear (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes